CLINICAL TRIAL: NCT00421239
Title: Retrospective Study of Hypertensive Urgencies in Patients With Arterial Hypertension
Brief Title: Risk Factors of Hypertensive Urgencies
Acronym: OSADA
Status: Completed | Type: Observational
Sponsor: Russian Cardiology Research and Production Center (Other)
Collaborators: KRKA (Industry)
Responsible Party: VNOK, Society of Cardiology of the Russian Federation
Other Study IDs: NCT00421239
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Hypertensive Urgency
Keywords: hypertensive urgency; arterial hypertension
MeSH Terms: conditions — Hypertensive Crisis; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
- B

SUMMARY:
The purpose of this study is to determine whether frequent hypertensive urgencies increase the risk of cardiovascular events in patients with arterial hypertension.

DETAILED DESCRIPTION:
The spectrum of disorders associated with arterial hypertension (AH) encompasses chronic uncomplicated hypertension and the hypertensive crises, including hypertensive urgences and emergencies. Hypertensive crises accounted for more than 25% of all patient visits to a medical section of an emergency department, with hypertensive urgences (HU) accounting for two-third of these cases. Hypertensive crises, without prompt treatment, are often associated with morbidity and mortality. We propose to conduct a population-based case-control study of HU in areas of the Russian Federation. We will include about thirty study centers and one data coordinating center and will recruit study participants over a period of one years. We plan to conduct in-person interviews with 1,500 cases and 1,500 controls to elicit information on demographic background and history of exposures. We intend to test about 20-25 risk factors of HU thus calculated target number of subject is 3000 pts. We're going to get access to hospital lists in each study center. From the database we'll select patients with AH and recruit every third participant who came to hospital or/and policlinic. Every selected participant will be asked to respond to some questions by phone and be divided into two groups. Participants who have HU two weeks before the call will be questioned about level of arterial pressure and treatment during HU. Participants with often HU (every week or more) will be included into first group (prevalent cases, group A). Participants with seldom HU (every month or less) will be included into second group (controls, group B). Cases and controls will be selected from the same population of AH patients. Questionnaire contains information about age, gender, tobacco use, data about HU (frequency, treatment and its complications), antihypertensive and concomitant treatment, level of blood pressure, regularity of taking antihypertensive drugs, associated clinical conditions (cerebrovascular disease, heart disease, renal disease, peripheral vascular disease), PCI, CABG, if it be possible we intend to collect information of factors influencing prognosis (fasting plasma glucose, dyslipidaemia, serum creatinine, serum uric acid, left ventricular hypertrophy).

ELIGIBILITY:
Inclusion Criteria:

* Cases: every third patient from hospital/policlinic database who are diagnosed with arterial hypertension (SBP/DBP>140/90 Hg or taking anti hypertensive drugs) and with frequent (weekly or daily) hypertensive urgencies (SBP/DBP≥180/110 Hg) will be potentially eligible for the study.
* Controls will be selected from the same population of participants by random telephone dialing to every third patient with arterial hypertension (SBP/DBP>140/90 Hg or taking anti hypertensive drugs) and with seldom (monthly, several times in the year or never) hypertensive urgencies.

Exclusion Criteria:

* Hypertensive emergency

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from hospital/policlinic database by random telephone dialing to every third patient who are diagnosed with arterial hypertension (SBP/DBP>140/90 Hg or taking antihypertensive drugs)
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2007-01; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evgeniy I Chazov, MD, Study Chair — Russian Cardiology Research and Production Center
Locations (1):
- Russian Cardiology Research and Production Center, Moscow, Russia